CLINICAL TRIAL: NCT04882098
Title: A Phase 3b, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Subcutaneously Administered Guselkumab in Improving the Signs and Symptoms and Inhibiting Radiographic Progression in Participants With Active Psoriatic Arthritis
Brief Title: A Study of Guselkumab in Participants With Active Psoriatic Arthritis
Acronym: APEX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108957; CNTO1959PSA3004 (Other: Janssen Research & Development, LLC); 2020-004981-20 (EudraCT Number); 2023-504734-21-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab and Placebo (Experimental): Participants will receive guselkumab and placebo subcutaneously (SC) to maintain the blind. Participants who have not discontinued will be eligible to enter a long-term extension (LTE) and will receive guselkumab and placebo SC. After the study is unblinded to the investigative sites, participants will receive guselkumab and no longer be required to dose with placebo to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab SC. Participants who have not discontinued will be eligible to enter an LTE and will receive guselkumab SC.
  Interventions: Drug: Guselkumab
- Group 3: Placebo Followed by Guselkumab (Experimental): Participants will receive placebo SC and will cross over to receive SC guselkumab. Participants who have not discontinued will be eligible to enter an LTE and will receive guselkumab SC.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive guselkumab as SC injection.
  Other Names: CNTO 1959
Drug: Placebo — Participants will receive matching placebo as SC injection.
  Arms: Group 1: Guselkumab and Placebo; Group 3: Placebo Followed by Guselkumab

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab treatment in participants with active psoriatic arthritis (PsA) by assessing the reduction in signs and symptoms of PsA.

ELIGIBILITY:
Inclusion Criteria:

* Have active psoriatic arthritis (PsA) despite previous non-biologic disease-modifying antirheumatic drug (DMARD), apremilast, and/or nonsteroidal anti-inflammatory drug (NSAID) therapy
* Have a diagnosis of PsA for at least 6 months before the first administration of study agent and meet Classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by: at least 3 swollen joints and 3 tender joints at screening and at baseline; and C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligrams per deciliter (mg/dL) at screening from the central laboratory
* Have >= 2 joints with erosions on baseline radiographs of the hands and feet as determined by central read
* Have at least one of the following PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis, with at least one psoriatic plaque of >= 2 centimeter (cm) diameter or nail changes consistent with psoriasis

Exclusion Criteria:

* Has known allergies, hypersensitivity, or intolerance to study intervention or its excipients
* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy, including but not limited to rheumatoid arthritis (RA), axial spondyloarthritis (AS)/non-radiographic axial spondyloarthritis (nr-axSpA), systemic lupus erythematosus, or Lyme disease
* Has previously received any biologic treatment
* Has ever received tofacitinib, baricitinib, filgotinib, peficitinib, decernotinib, upadacitinib or any other Janus kinase (JAK) inhibitor
* Has received any systemic immunosuppressants (example, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1054 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2027-10-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (274):
- United States (23):
  - Rheumatology Associates, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Research PLLC, Flagstaff, Arizona
  - Arizona Arthritis & Rheumatology Associates PC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Tucson, Arizona
  - Advanced Medical Research, La Palma, California
  - Rheumatology Center of San Diego, San Diego, California
  - Medvin Clinical Research, Inc., Whittier, California
  - Heuer M.D. Research, Orlando, Florida
  - The Arthritis Center, Inc., Palm Harbor, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Klein And Associates M D P A, Hagerstown, Maryland
  - Advanced Rheumatology, Lansing, Michigan
  - Arthritis Consultants, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - PMG Research of Salisbury, Salisbury, North Carolina
  - STAT Research, Inc., Springboro, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Dr. Ramesh Gupta, Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Adriana Pop Moody MD Clinic PA, Corpus Christi, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Arthritis And Osteoporosis Clinic, Waco, Texas
- Australia (5):
  - The Queen Elizabeth Hospital, Adelaide
  - Southern Clinical Research, Hobart
  - Emeritus Research, Melbourne
  - Eastern Health - Box Hill Hospital, Melbourne
  - Rheumatology Research Unit, Sunshine Coast
- Bosnia and Herzegovina (4):
  - University Clinical center Republic of Srpska, Banja Luka
  - Health center Gradiska, Gradiška
  - Clinical hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Sarajevo
- Bulgaria (13):
  - UMHAT Kaspela, Plovdiv
  - MHAT Trimantium, Plovdiv
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Multiprofile Hosptal for Active Treatment Eurohospital Plovdiv, Plovdiv
  - Medical Center Unimed Plovdiv, Plovdiv
  - Medical Center Teodora, Rousse
  - Medical Center Medconsult-Pleven, Sevlievo
  - UMHAT Sv. Ivan Rilski, Sofia
  - UMHAT St. Ivan Rilski, Sofia
  - DCC XVII-Sofia EOOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - St Ivan Rilski University Multiprofile Hospital For Active Treatment, Sofia
  - DCC Convex EOOD, Sofia
- Canada (4):
  - Eastern Regional Health Authority St Clares Mercy Hospital, St. John's, Newfoundland and Labrador
  - Toronto Western Hospital, Toronto, Ontario
  - Group De Recherche En Rhumatologie Et Maladies Osseuses, Québec, Quebec
  - Centre de Recherche Musculo Squelettique, Trois-Rivières, Quebec
- China (24):
  - Affiliated Hospital of Hebei University, Baoding
  - The First Affiliated Hospital of Baotou Medical University, Baotou
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Bethune Hospital of Jilin University, Changchun
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - the 3rd Affiliated Hospital,Sun Yansen University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Linyi City People Hospital, Linyi
  - The First Affiliated Hospital of NanChang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Pingxiang People's Hospital, Pingxiang
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai skin disease hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - The hospital of Shanxi Universtidy, Taiyuan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Croatia (6):
  - Ch Osijek, Osijek
  - KBC Rijeka, Rijeka
  - University Hospital Center Split, Split
  - Klinicki bolnicki centar Zagreb, Zagreb
  - Medicinski centar Kuna & Peric, Zagreb
  - University Hospital Sveti Duh, Zagreb
- Czechia (14):
  - Revmaclinic, Brno
  - Revmatologie s r o, Brno
  - Revmacentrum MUDr Mostera s r o, Brno-Židenice
  - L K N Arthrocentrum, Hlučín
  - CCBR Ostrava s r o, Ostrava
  - MUDr Rosypalova s r o, Ostrava
  - CCBR Klinicka centra Czech, a.s., Pardubice
  - Revmatologicky institut, Prague
  - CCR Prague s.r.o., Prague
  - Revmatologicka ambulance, Prague
  - Affidea Praha s r o, Prague
  - Fakultni nemocnice v Motole, Prague
  - Medical Plus S R O, Uherské Hradiště
  - PV Medical S R O, Zlín
- Estonia (3):
  - OU Innomedica, Tallinn
  - North Estonia Medical Centre, Tallinn
  - Sihtasutus Tartu Ulikooli Kliinikum - Nahahaiguste Kliinik, Tartu
- Georgia (11):
  - LTD Unimed Adjara, Batumi
  - LTD Clinic LJ, Kutaisi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - Raymann Ltd, Tbilisi
  - J S C K Eristavi National Cen, Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd, Tbilisi
  - LTD MediClub Georgia, Tbilisi
  - Consilium Medulla-multiprofile clinic Ltd, Tbilisi
  - Ltd Medicore, Tbilisi
  - JSC Evex Hospitals, Tbilisi
  - LTD The First Medical Center, Tbilisi
- Germany (7):
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Praxis fur Klinische Studien und Praxis fur Orthopadie, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Institut Fur Praventive Medizin Klinische Forschung GbR, Magdeburg
  - Gemeinschaftspraxis Dres. Quist, Mainz
  - Rheumazentrum Ratingen, Ratingen
- Greece (5):
  - Naval Hospital of Athens, Athens
  - Hippokration Hospital, Athens
  - Laiko General Hospital of Athens, Athens
  - University Hospital Of Larissa, Biopolis, Larissa
  - Democritus University of Thrace, Xánthi
- Hungary (11):
  - Revita Rendelo, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Uno Medical Trials Ltd., Budapest
  - Qualiclinic Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Synexus Magyarorszag Kft, Gyula
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szegedi Tudományegyetem, ÁOK, Szent-Györgyi Albert Klinikai Központ, Szeged
  - Csongrád Megyei Dr. Bugyi István Kórház, Szentes
  - MAV Korhaz es Rendelointezet, Szolnok
  - Synexus Magyarorszag Kft, Zalaegerszeg
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - PO G.Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania
  - Ospedale San Raffaele, IRCCS, Milan
  - AOU Università degli Studi della Campania L. Vanvitelli, Napoli
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Università di Roma La Sapienza, Roma
  - Complesso Integrato Columbus, Rome
  - A.O.U. Città della Salute e della Scienza, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Latvia (6):
  - M & M Centrs Ltd, Ādaži
  - P. Stradina Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
  - Riga 1st Hospital, Riga
  - J Kisis Ltd, Riga
  - Orto Clinic Ltd, Riga
- Lithuania (5):
  - Practice Dr Pociene Gilvina, Kaunas
  - Lietuvos sveikatos mokslų universiteto ligoninė Kauno klinik, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - JSC Inlita, Santaros KTC, Vilnius
- Malaysia (6):
  - Hospital Selayang, Batu Caves
  - Hospital Raja Permaisuri Bainun, Ipoh
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Melaka, Malacca
  - Sunway Medical Centre, Petaling Jaya
  - Hospital Tuanku Jaafar, Seremban
- Philippines (9):
  - Angeles University Foundation Medical Center, Angeles
  - Cebu Doctors' University Hospital, Cebu
  - De La Salle University Medical Center, Dasmariñas
  - Southern Philippines Medical Center, Davao City
  - Davao Doctors Hospital, Davao City
  - University of Perpetual Help Dalta Medical Center, Inc, Las Piñas
  - Manila Doctors Hospital, Manila
  - Medical Center Manila, Manila
  - Philippine General Hospital, Manila
- Poland (17):
  - Osteo-Medic s.c A. Racewicz, J Supronik, Bialystok
  - ClinicMed Badurski i Wspolnicy Spolka Jawna, Bialystok
  - Nasz Lekarz Przychodnie Medyczne, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Ambulatorium Barbara Bazela, Elblag
  - Medica Pro Familia sp z o o S K A, Gdynia
  - Pratia MCM Krakow, Krakow
  - REUMED Zespol Poradni Specjalistycznych Filia nr 2, Lublin
  - NZOZ Lecznica Mak-Med sc, Nadarzyn
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Prywatna Praktyka Lekarska Prof Um Dr Hab Med Pawel Hrycaj, Poznan
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Medycyna Kliniczna, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Reumatika-Centrum Reumatologii, NZOZ, Warsaw
  - DERMMEDICA Sp.z o.o., Wroclaw
- Russia (22):
  - Chelyabinsk Regional Clinical Dermatovenerological Dispensary, Chelyabinsk
  - LLC Aliance Biomedical-Ural group, Izhevsk
  - State Budgetary Educational Institution of High Professional Education, Kazan'
  - Medical Center LLC Maxsimum Zdoroviya, Kemerovo
  - LLC Family Outpatient Clinic # 4, Moscow
  - GUZ of Moscow City Clinical Hospital # 1 n.a.N.I.Pirogov, Moscow
  - GU Moscow Regional Research Clinical Institute n.a. M.F.Vla, Moscow
  - FGBU Research Institute of Rheumatology named V.A.Nasonova, Moscow
  - LLC Consultative and Diagnostic Center of Rheumatology Heal, Novosibirsk
  - GBUZ Orenburg Clinical Regional Hospital, Orenburg
  - Republican Hospital n.a.V.A.Baranov, Petrozavodsk
  - Ryazan Regional Clinical Dermatovenerological Dispensary, Ryazan
  - Ryazan Regional Clinical Cardiology Center, Ryazan
  - Ryazan Regional Clinical Hospital, Ryazan
  - Northen-Western State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - Federal North-West Medical Research Centre, Saint Petersburg
  - LLC Sanavita, Saint Petersburg
  - Sararov Regional Clinical Hospital, Saratov
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - State Budget Healthcare Institution of Vladimir Region Regional Clinical Hospital, Vladimir
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
  - Clinical Hospital #3, Yaroslavl
- Serbia (5):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Special Hospital for Rheumatic Diseases, Novi Sad
- Slovakia (4):
  - Paediatric University Hospital, Košice
  - Reumatologicka ambulancia, Martin
  - Chiremed, s.r.o., Púchov
  - Reumex s.r.o, Rimavská Sobota
- Slovenia (3):
  - Splosna bolnisnica Izola, Izo
  - Bolnica Dr. Petra Drzaja, Ljubljana
  - UKC Maribor Dermatology clinic, Maribor
- South Korea (7):
  - Soonchunhyang University Cheonan Hospital, Cheonan-si
  - Chonnam National University Hospital, Gwangju
  - Hanyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (12):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. de Mostoles, Móstoles
  - Hosp. Univ. Virgen de La Arrixaca, Murcia
  - Hosp. Univ. Infanta Sofia, San Sebastián de los Reyes
  - Complejo Hospitalario Universitario de Santiago. Servicio de Aparato Digestivo, Santiago de Compostela
  - Hosp. Nuestra Senora de La Esperanza, Santiago de Compostela
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Infanta Luisa, Seville
- Taiwan (8):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
  - Chi Mei Medical Center Yong Kang, Yung-Kang
- Turkey (Türkiye) (4):
  - Akdeniz University Medical Faculty, Istanbul
  - Izmir Katip Celebi University, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Selcuk University Medical Faculty, Konya
- Ukraine (21):
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Derzhavna ustanova Natsionalnyi instytut terapii imeni L.T.Maloi NAMN Ukrainy viddil klinichnoi, Kharkiv
  - Municipal Institution Regional hospital-center of emergency care and disasters medicine, Kharkiv
  - Khmelnitska oblasna likarnia, Khmelnitsky
  - TOV Revmocentr, Kiev
  - Komunalnyi zaklad Kryvorizka miska klinichna likarnia #2 Dnipropetrovskoi oblasnoi rady, Kryvyi Rih
  - Medical Research and Practice Center Medbud of the Public Joint Stock Holding Company Kyivmiskbud, Kyiv
  - State Institution Railway clinical Hospital 2, Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - Olexandrivska Clinical Hospital of Kyiv City, Kyiv
  - Kyivska oblasna klinichna likarnia, Kyiv
  - Center of Family Medicine Plus LLC, Kyiv
  - Kyiv Railway Station Clinical Hospital #2, Kyiv
  - Odeska oblasna klinichna likarnia, Odesa
  - Multidisciplinary Medical Center of Odessa National Medical University, Odesa
  - ME Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of Poltava Regional Consuil, Poltava
  - Sumska oblasna klinichna likarnia, Sumy
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
  - Medical Center LTD Health Clinic Department of Cardiology and Rheumatology, Vinnytsia
  - Naukovo-doslidnyi inst. Reabilit. Pyrogova [Revmatologichne], Vinnytsia
  - Zhytomyr Central City Hospital #1, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Ritchlin CT, Coates LC, Mease PJ, van der Heijde D, Song J, Jiang Y, Shawi M, Kollmeier AP, Rahman P. The effect of guselkumab on inhibiting radiographic progression in patients with active psoriatic arthritis: study protocol for APEX, a Phase 3b, multicenter, randomized, double-blind, placebo-controlled trial. Trials. 2023 Jan 10;24(1):22. doi: 10.1186/s13063-022-06945-y. PMID 36627711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1054 participants were randomized, and all received study drug and were analyzed for safety (Safety Analysis Set). 5 Ukrainian sites were excluded from the main efficacy analysis (Modified FAS, N=1020), as they were unable to support key study operations due to the crisis in Ukraine and neighboring countries/territories beginning 2022-02-24. Results are currently reported until the primary completion date (30 December 2024). Results of remaining duration will be reported upon study completion.
Groups:
- Group 1: Guselkumab 100 mg q8w: Participants received guselkumab 100 milligram (mg) subcutaneous (SC) injection at Weeks 0 and 4, then every 8 weeks (q8w) starting from Week 12 through Week 44 and placebo matched to guselkumab SC injections q8w starting from Week 8 through Week 48 to maintain the blind. After the Week 48 database lock and subsequent full unblinding, placebo injections were no longer required. At Week 48, eligible participants had the option to enter a long-term extension (LTE) and continued to receive guselkumab 100 mg SC injection every 4 weeks (q4w) up to Week 156 and then followed up for safety until Week 168. Participants who did not enter LTE at Week 48 were followed up for safety till Week 60.
- Group 2: Guselkumab 100 mg q4w: Participants received guselkumab 100 mg SC injections q4w from Week 0 through Week 48. At Week 48, eligible participants had the option to enter a LTE and continued to receive guselkumab 100 mg SC injection q4w up to Week 156 and then followed up for safety until Week 168. Participants who did not enter LTE at Week 48 were followed up for safety till Week 60.
- Group 3: Placebo Followed by Guselkumab: Participants received placebo matched to guselkumab SC injections q4w starting from Week 0 through Week 20. Participants then crossed over and received guselkumab 100 mg SC injections q4w from Week 24 through Week 48. At Week 48, eligible participants had the option to enter a LTE and continued to receive guselkumab 100 mg SC injection q4w up to Week 156 and then followed up for safety until Week 168. Participants who did not enter LTE at Week 48 were followed up for safety till Week 60.
Period: Overall Study
Arm/Group | Group 1: Guselkumab 100 mg q8w | Group 2: Guselkumab 100 mg q4w | Group 3: Placebo Followed by Guselkumab
Started | 388 | 280 | 386
Modified Full Analysis Set (Modified full analysis set included all participants who were randomized, excluding participants from Ukrainian sites rendered unable to support key study operations due to major disruption.) | 371 | 273 | 376
Completed | 370 | 270 | 372
Not Completed | 18 | 10 | 14
Not completed — Adverse Event | 7 | 2 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 9
Not completed — Subject refused further study treatment | 1 | 0 | 0
Not completed — Other | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Guselkumab 100 mg q8w: Participants received guselkumab 100 mg SC injection at Weeks 0 and 4, then q8w starting from Week 12 through Week 44 and placebo matched to guselkumab SC injections q8w starting from Week 8 through Week 48 to maintain the blind. After the Week 48 database lock and subsequent full unblinding, placebo injections were no longer required. At Week 48, eligible participants had the option to enter a LTE and continued to receive guselkumab 100 mg SC injection every q4w up to Week 156 and then followed up for safety until Week 168. Participants who did not enter LTE at Week 48 were followed up for safety till Week 60.
- Total: Total of all reporting groups
Arm/Group | Group 1: Guselkumab 100 mg q8w | Group 2: Guselkumab 100 mg q4w | Group 3: Placebo Followed by Guselkumab | Total
Number analyzed (Participants) | 388 | 280 | 386 | 1054
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.03) | 52.3 (13.15) | 53.4 (12.92) | 52.9 (13.02)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 311 | 229 | 304 | 844
  From 65 to 84 years | 77 | 51 | 82 | 210
  85 years and over | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 127 | 170 | 479
  Male | 206 | 153 | 216 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 8 | 18
  Not Hispanic or Latino | 382 | 276 | 378 | 1036
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 61 | 38 | 61 | 160
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 0 | 4
  Black or African American | 2 | 0 | 0 | 2
  White | 322 | 240 | 321 | 883
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 3 | 3 | 9
  Bosnia and Herzegovina | 24 | 13 | 25 | 62
  Bulgaria | 32 | 28 | 35 | 95
  Canada | 3 | 1 | 1 | 5
  China | 25 | 17 | 27 | 69
  Croatia | 8 | 2 | 5 | 15
  Estonia | 3 | 2 | 5 | 10
  Georgia | 37 | 30 | 33 | 100
  Germany | 4 | 1 | 0 | 5
  Greece | 1 | 0 | 1 | 2
  Hungary | 5 | 10 | 10 | 25
  Israel | 6 | 2 | 7 | 15
  Italy | 3 | 2 | 2 | 7
  Latvia | 13 | 4 | 4 | 21
  Lithuania | 16 | 15 | 23 | 54
  Malaysia | 4 | 2 | 5 | 11
  Philippines | 32 | 18 | 23 | 73
  Poland | 38 | 25 | 27 | 90
  Russian Federation | 20 | 16 | 19 | 55
  Serbia | 27 | 20 | 28 | 75
  Slovakia | 6 | 6 | 6 | 18
  Slovenia | 1 | 1 | 0 | 2
  Korea, South | 0 | 0 | 1 | 1
  Spain | 9 | 9 | 14 | 32
  Taiwan | 1 | 1 | 3 | 5
  Turkey | 1 | 0 | 1 | 2
  Ukraine | 35 | 25 | 39 | 99
  United States | 10 | 11 | 13 | 34
  Czech Republic | 21 | 16 | 26 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR 20 response: >=20% improvement from baseline (bl) in both swollen (66 joints), tender (68 joints) joint count, >=20% improvement from bl in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100mm, 0=no pain, 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100mm, 0=excellent, 100=poor), physician's global assessment of disease activity (VAS; 0-100mm, 0=no arthritis activity,100=extremely active arthritis), HAQ-DI (questionnaire assessing 8 functional areas; 0-3, 0=no difficulty, 3=inability to perform task in area), and CRP. Natural Disaster (ND)-site inaccessible due to COVID-19. Major Disruption (MD)-disruption involving Ukraine and neighboring countries/territories. Intercurrent event (ICE) handling: Composite-discontinue study drug not due to ND/MD, initiate/increase DMARD/oral corticosteroid, initiate prohibited PsA treatment; Hypothetical-discontinue/severe noncompliance of study drug due to ND/MD.
Time Frame: At Week 24
Population: Analysis population is Modified FAS (mFAS). Participants who achieved ACR 20 response at Week 24 and did not meet any Composite Strategy ICEs before Week 24 were considered as responders. Participants who met any Composite Strategy ICEs before Week 24 were considered non-responders. Participants who met Hypothetical Strategy ICEs, or missed data due to ND/MD, had affected visits imputed using multiple imputation. Other missing data were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Guselkumab 100 mg q8w | Group 2: Guselkumab 100 mg q4w | Group 3: Placebo Followed by Guselkumab
Number analyzed (Participants) | 371 | 273 | 376
percentage of participants | 68.3 | 66.6 | 47.0
Statistical Analysis 1: Comparison: Group 1: Guselkumab 100 mg q8w vs Group 3: Placebo Followed by Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 21.3, 95% CI 2-sided [14.4 to 28.2]
Statistical Analysis 2: Comparison: Group 2: Guselkumab 100 mg q4w vs Group 3: Placebo Followed by Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 19.7, 95% CI 2-sided [12.1 to 27.2]

2. Secondary Outcome: Change From Baseline in Psoriatic Arthritis (PsA) Modified Van Der Heijde-Sharp (vdH-S) Total Score at Week 24
Description: Modified vdH-S score was sum of erosion score (hand, feet) and joint space narrowing (JSN) score (hand, feet). Joint erosion score was total erosion severity in 40 joints of 2 hands and 12 joints of 2 feet, maximum erosion score=320. Each hand joint was scored on 0 to 5 with 0 =no erosion, 5 =complete collapse of bone. Foot joint was scored on 0 to 10, 0 =no erosion, 10 =complete collapse of bone. JSN score was total JSN score in same 52 joints, each joint scored on 0 to 4 with 0 indicating no JSN, and 4 indicating absence of joint space, maximum JSN score=208. Maximum modified vdH-S score=528. Higher score =severe structural destruction and complete loss of joint spaces. Natural Disaster (ND)-site inaccessible due to COVID-19. Major Disruption (MD)-disruption involving Ukraine and neighboring countries/territories. Intercurrent event (ICE) handling: Hypothetical-discontinue/severe noncompliance of study drug due to ND/MD
Time Frame: Baseline (after first administration of study drug) and Week 24
Population: Modified full analysis set included all participants who were randomized, excluding participants from Ukrainian sites rendered unable to support key study operations due to major disruption. Participants who met Hypothetical Strategy ICEs had affected visits imputed using multiple imputation. Missing data were also imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Group 1: Guselkumab 100 mg q8w | Group 2: Guselkumab 100 mg q4w | Group 3: Placebo Followed by Guselkumab
Number analyzed (Participants) | 371 | 273 | 376
Score on a scale | 0.54 [0.14 to 0.95] | 0.55 [0.10 to 1.00] | 1.35 [0.94 to 1.75]
Statistical Analysis 1: Comparison: Group 1: Guselkumab 100 mg q8w vs Group 3: Placebo Followed by Guselkumab; Test type: Superiority; p < 0.001, ANCOVA; Least Square Mean Difference = -0.8, 95% CI 2-sided [-1.28 to -0.33]
Statistical Analysis 2: Comparison: Group 2: Guselkumab 100 mg q4w vs Group 3: Placebo Followed by Guselkumab; Test type: Superiority; p = 0.002, ANCOVA; Least Square Mean Difference = -0.8, 95% CI 2-sided [-1.31 to -0.28]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

5. Secondary Outcome: Number of Participants With Reasonably Related Adverse Events (AEs)
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

6. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation of Study Intervention
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

7. Secondary Outcome: Number of Participants With Treatment Emergent Infections
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

8. Secondary Outcome: Number of Participants With Injection-site Reactions Leading to Discontinuation of Study Intervention
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

9. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

10. Secondary Outcome: Number of Participants With Maximum Common Terminology Criteria for Adverse Events (CTCAE) Toxicity Grade Laboratory Values
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

11. Secondary Outcome: Serum Guselkumab Concentration
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

12. Secondary Outcome: Number of Participants With Anti-guselkumab Antibodies
Time Frame: From baseline (after first administration of study drug) up to 168 weeks
Reporting Status: Not Posted, anticipated posting 2029-12

ADVERSE EVENTS:
Time Frame: All cause mortality, SAEs, and non-SAEs: From baseline (after first administration of study drug) up to 24 weeks.
Description: Safety analysis set included all participants who received at least one (complete or partial) administration of study intervention, that is, the treated population.
Arm/Group | Group 1: Guselkumab 100 mg q8w | Group 2: Guselkumab 100 mg q4w | Group 3: Placebo Followed by Guselkumab
All-Cause Mortality (participants affected / at risk) | 0/388 | 1/280 | 0/386
Serious Adverse Events (participants affected / at risk) | 12/388 | 5/280 | 10/386
Other Adverse Events (participants affected / at risk) | 41/388 | 22/280 | 42/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Guselkumab 100 mg q8w (N=388) | Group 2: Guselkumab 100 mg q4w (N=280) | Group 3: Placebo Followed by Guselkumab (N=386)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 1
Covid-19 Pneumonia (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Superficial Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Guselkumab 100 mg q8w (N=388) | Group 2: Guselkumab 100 mg q4w (N=280) | Group 3: Placebo Followed by Guselkumab (N=386)
Covid-19 (Infections and infestations) | 22 | 8 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 20 | 15 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT04882098/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04882098/SAP_001.pdf